CLINICAL TRIAL: NCT00707031
Title: A Randomized, Open-label, Active-controlled, 2-arm Parallel-group, Multicenter 24-week Study Followed by an Extension Assessing the Efficacy and Safety of AVE0010 Versus Exenatide on Top of Metformin in Patients With Type 2 Diabetes Not Adequately Controlled With Metformin
Brief Title: GLP-1 Receptor Agonist Lixisenatide Versus Exenatide in Patients With Type 2 Diabetes for Glycemic Control and Safety Evaluation, on Top of Metformin
Acronym: GETGOAL-X
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6019; 2007-005883-28 (EudraCT Number)
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: hyperglycemia, GLP-1, metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — lixisenatide; Exenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide (Experimental): 2-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Metformin
- Exenatide (Active Comparator): 1-step initiation regimen of exenatide: 5 mcg twice daily (BID) for 4 weeks, followed by 10 mcg BID up to the end of treatment.
  Interventions: Drug: Exenatide; Device: Prefilled pen injector; Drug: Metformin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Lixisenatide
Device: Pen auto-injector
  Other Names: OptiClik®
  Arms: Lixisenatide
Drug: Exenatide — Self administered by subcutaneous injections twice daily within the hour preceding breakfast and within the hour preceding dinner.
  Other Names: Byetta®
  Arms: Exenatide
Device: Prefilled pen injector
  Arms: Exenatide
Drug: Metformin — Metformin to be continued at stable dose (at least 1.5 gram per day) up to the end of treatment.

SUMMARY:
The purpose of this study is to compare the benefits and risks of lixisenatide (AVE0010) in comparison to exenatide (Byetta®), as an add-on treatment to metformin, over a period of 24 weeks of treatment, followed by an extension.

The primary objective is to assess the effects of lixisenatide in comparison to exenatide (Byetta®), as an add-on treatment to metformin, on glycemic control in terms of glycosylated hemoglobin (HbA1c) reduction (absolute change) at Week 24.

The secondary objectives are to assess the effects of lixisenatide on percentage of patients reaching HbA1c less than 7 percent (%) or HbA1c less than or equal to (<=) 6.5%, fasting plasma glucose (FPG), body weight; to evaluate safety, tolerability and to assess the impact of gastrointestinal tolerance on quality of life (QoL) (patient assessment of upper gastrointestinal disorders - quality of life [PAGI-QOL]).

DETAILED DESCRIPTION:
Patients who complete the 24-week main open-label treatment would undergo a variable open-label extension treatment, which ends for all patients at approximately the scheduled date of Week 76 visit (Visit 24) for the last randomized patient.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed for at least 1 year before screening visit, insufficiently controlled with metformin at a stable dose of at least 1.5 gram per day for at least 3 months prior to screening visit

Exclusion Criteria:

* HbA1c less than (<) 7% or greater than (>) 10% at screening
* At the time of screening age < legal age of majority
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* Type 1 diabetes mellitus
* Treatment with another antidiabetic pharmacological agent than metformin within the 3 months preceding the screening
* FPG at screening >250 milligram per deciliter (mg/dL) (13.9 millimole per liter [mmol/L])
* Body mass index (BMI) less than or equal to (<=) 20 kilogram per square meter (kg/m^2)
* Weight change of >5 kg during the 3 months preceding the study
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease
* History of metabolic acidosis, including diabetic ketoacidosis, within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within 3 months prior to the time of screening
* Within the last 6 months prior to screening, history of myocardial infarction, stroke, or heart failure requiring hospitalization
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic blood pressure or diastolic blood pressure >180 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Laboratory findings at the time of screening: aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase: >2 times upper limit of the normal (ULN) laboratory range; amylase and/or lipase: >3 times ULN; total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome); hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100 000/ mm^3; positive test for Hepatitis B surface antigen and/or Hepatitis C antibody; and positive serum pregnancy test in females of childbearing potential
* Any clinically significant abnormality identified on physical examination, laboratory tests, electrocardiogram or vital signs at the time of screening that, in the judgment of the investigator or any sub-investigator, precludes safe completion of the study or constrains efficacy assessment
* Patients who are considered by the investigator or any sub-investigator as inappropriate for this study for any reason (for example, impossibility to meet specific protocol requirements, such as attending scheduled visits, being able to do self-injections; likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol; investigator or any sub-investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol)
* Use of other oral or injectable antidiabetic or hypoglycemic agents than metformin (for example, sulfonylurea, alpha-glucosidase inhibitor, thiazolidinedione, rimonabant, exenatide, dipeptidyl-peptidase-4 inhibitors, insulin) within 3 months prior to the time of screening
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to the time of screening
* Use of any investigational drug within 3 months prior to study
* Participation in any previous study with lixisenatide
* Renal impairment defined with serum creatinine >1.4 mg/dL in women and serum creatinine >1.5 mg/dL in men
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to, gastroparesis and gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening
* Allergic reaction to any glucagon like peptide-1 (GLP-1) agonist in the past (for example, exenatide, liraglutide) or to metacresol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (18):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, San Juan, Puerto Rico
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden

REFERENCES:
- [Result] Rosenstock J, Raccah D, Koranyi L, Maffei L, Boka G, Miossec P, Gerich JE. Efficacy and safety of lixisenatide once daily versus exenatide twice daily in type 2 diabetes inadequately controlled on metformin: a 24-week, randomized, open-label, active-controlled study (GetGoal-X). Diabetes Care. 2013 Oct;36(10):2945-51. doi: 10.2337/dc12-2709. Epub 2013 May 22. PMID 23698396
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 122 centers in 18 countries between June 23, 2008 and November 18, 2010. The overall duration of treatment was at least 76 weeks (24 weeks main open-label treatment; variable open-label extension treatment).
Pre-assignment Details: A total of 1243 patients were screened of which 604 were screen failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7% and less than or equal to 10%). A total of 639 patients were randomized.
Groups:
- Lixisenatide: 2-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Exenatide: 1-step initiation regimen of exenatide: 5 mcg twice daily (BID) subcutaneously for 4 weeks, followed by 10 mcg BID up to the end of treatment.
Period: Overall Study
Arm/Group | Lixisenatide | Exenatide
Started | 320 (Randomized) | 319
Treated/Safety Population | 318 (All patients who received at least 1 dose, regardless of amount of treatment administered.) | 316
Modified Intent-to-Treat Population | 315 (All patients who received at least 1 dose;had baseline;at least 1 post-baseline efficacy assessment.) | 315
Completed | 216 | 220
Not Completed | 104 | 99
Not completed — Adverse Event | 45 | 45
Not completed — Lack of Efficacy | 19 | 6
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Poor Compliance to Protocol | 7 | 13
Not completed — Familial or Personal Reasons | 12 | 15
Not completed — Serious Noncompliance | 2 | 3
Not completed — Sponsor Decision | 9 | 8

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who received at least 1 dose of study drug, regardless of the amount of treatment administered. In addition, 5 patients from one site with serious noncompliance issues were excluded from all analysis populations.
Groups:
- Lixisenatide: 2-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Exenatide: 1-step initiation regimen of exenatide: 5 mcg BID subcutaneously for 4 weeks, followed by 10 mcg BID up to the end of treatment.
- Total: Total of all reporting groups
Arm/Group | Lixisenatide | Exenatide | Total
Number analyzed (Participants) | 318 | 316 | 634
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (9.2) | 57.6 (10.7) | 57.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 129 | 296
  Male | 151 | 187 | 338
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian/White | 296 | 292 | 588
  Race: Black | 8 | 10 | 18
  Race: Asian/Oriental | 3 | 4 | 7
  Race: Other | 11 | 10 | 21
  Ethnicity: Hispanic | 87 | 83 | 170
  Ethnicity: Non Hispanic | 231 | 233 | 464
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 7.95 (0.81) | 7.97 (0.78) | 7.96 (0.80)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 9.7 (2.0) | 9.7 (2.3) | 9.7 (2.1)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 94.0 (19.6) | 96.1 (22.5) | 95.0 (21.13)
Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QOL) Total Score [Mean (Standard Deviation); unit: units on a scale] — A 30-item self-administered questionnaire to measure health related quality of life (QOL) of patients with upper gastrointestinal disorders during past 2 weeks; consisted of 5 dimensions (subscales). Each item rated on a 0-5 point Likert scale, where 0=none of the time and 5=all the time. Subscale score was calculated by dividing sum of all items of subscale by number of items in subscale. Total score was calculated by taking the mean of subscale scores. Subscale score and total score range from 0 to 5 with lower scores indicating better quality of life.
  units on a scale | 0.59 (0.7) | 0.56 (0.7) | 0.58 (0.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated by dividing body weight by the height squared.
  kilogram per square meter (kg/m^2) | 33.68 (6.27) | 33.51 (6.54) | 33.60 (6.40)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.78 (5.54) | 6.75 (4.87) | 6.76 (5.21)
Daily Metformin Dose [Mean (Standard Deviation); unit: milligram (mg)] | 2020.20 (459.41) | 2058.39 (453.23) | 2039.24 (456.38)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Absolute Change = HbA1c value at Week 24 minus HbA1c value at baseline. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 11 (Week 24) or Day 169 if Visit 11 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population:all randomized patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures. Last observation carried forward used. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- Lixisenatide: 2-step initiation regimen of lixisenatide.
- Exenatide: 1-step initiation regimen of exenatide.
Arm/Group | Lixisenatide | Exenatide
Number analyzed (Participants) | 295 | 297
percentage of hemoglobin | -0.79 (0.053) | -0.96 (0.054)
Statistical Analysis 1: Comparison: Lixisenatide vs Exenatide; To detect that upper confidence limit of 2-sided 95% confidence interval for least square (LS) mean difference between the 2 arms do not exceed 0.4% HbA1c, 300 patients per group would provide 96% power assuming a standard deviation of 1.3 and true difference in HbA1c between the 2 arms as 0; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the upper limit of the 2-sided 95% confidence interval of the difference between lixisenatide and exenatide on mITT population was <=0.4%; Statistical testing: 2-sided at significance level=0.05. Analysis of co-variance (ANCOVA) included treatment arms, randomization strata of screening HbA1c (<8.0, >=8.0%), BMI (<30, >=30 kg/m^2), country as fixed effects, baseline HbA1c as covariate; Least squares (LS) mean difference = 0.17, 95% CI 2-sided [0.033 to 0.297], Standard Error of Mean 0.067

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 1 day after the last dose of study drug, on or before Visit 11 (Week 24) or Day 169 if Visit 11 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using last observation carried forward (LOCF). Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide | Exenatide
Number analyzed (Participants) | 310 | 301
mmol/L | -1.22 (0.116) | -1.45 (0.119)

3. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 11 (Week 24) or Day 169 if Visit 11 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Lixisenatide | Exenatide
Number analyzed (Participants) | 295 | 296
kilogram | -2.96 (0.231) | -3.98 (0.232)

4. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 24
Description: The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 11 (Week 24) or Day 169 if Visit 11 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Exenatide
Number analyzed (Participants) | 295 | 297
percentage of participants | 48.5 | 49.8

5. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 24
Description: as for outcome 4
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Exenatide
Number analyzed (Participants) | 295 | 297
percentage of participants | 28.5 | 35.4

6. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During Main 24-Week Period
Description: Routine fasting self-monitored plasma glucose (SMPG) and central laboratory FPG (and HbA1c after week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after week 12) were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >270 milligram/deciliter (mg/dL) (15.0 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c > 8.5%. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Exenatide
Number analyzed (Participants) | 315 | 315
percentage of participants | 2.2 | 3.8

7. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 24
Description: as for outcome 4
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Groups:
- Exenatide: 2-step initiation regimen of exenatide.
Arm/Group | Lixisenatide | Exenatide
Number analyzed (Participants) | 295 | 296
percentage of participants | 25.1 | 31.4

8. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from hypoglycemia in which the patient required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration, for up to 116 weeks
Population: Safety population included all randomized patients who received at least 1 dose of study drug, regardless of the amount of treatment administered.
Measure: Number; unit: participants
Arm/Group | Lixisenatide | Exenatide
Number analyzed (Participants) | 318 | 316
participants
  Symptomatic Hypoglycemia | 16 | 46
  Severe Symptomatic Hypoglycemia | 0 | 0

9. Other Pre Specified Outcome: Quality of Life: Change From Baseline in Patient's Satisfaction to Treatment (PAGI-QOL) at Week 24
Description: PAGI-QOL: a 30-item self-administered questionnaire to measure health related QOL of patients with upper gastrointestinal disorders during past 2 weeks. Consists of 5 sub-scales. Each item rated on a 0-5 point Likert scale (0 [none of the time] to 5 [all the time]). Sub-scale score calculated by dividing sum of all items of subscale by number of items in the sub-scale. Total score calculated by taking mean of sub-scale scores. Sub-scale score and total score ranges from 0=none of the time (lowest score) to 5=all of the time (highest score) with lower scores indicating better QOL. The on-treatment period for this variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 11 (Week 24) or Day 169 if Visit 11 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline PAGI-QOL assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lixisenatide | Exenatide
Number analyzed (Participants) | 302 | 292
units on a scale | -0.09 (0.031) | -0.06 (0.032)

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration, for up to 116 weeks
Description: Median exposure to study treatment was 562 and 560 days in lixisenatide and exenatide treatment arms, respectively. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Arm/Group | Lixisenatide | Exenatide
Serious Adverse Events (participants affected / at risk) | 26/318 | 22/316
Other Adverse Events (participants affected / at risk) | 204/318 | 218/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (N=318) | Exenatide (N=316)
Appendicitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Retinopathy (Eye disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (N=318) | Exenatide (N=316)
Bronchitis (Infections and infestations) | 19 | 19
Influenza (Infections and infestations) | 29 | 32
Nasopharyngitis (Infections and infestations) | 49 | 35
Upper respiratory tract infection (Infections and infestations) | 18 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 18 | 48 — Hypoglycaemia adverse event is based on investigator reported hypoglycaemia.
Dizziness (Nervous system disorders) | 21 | 31
Headache (Nervous system disorders) | 46 | 31
Hypertension (Vascular disorders) | 19 | 10
Abdominal pain upper (Gastrointestinal disorders) | 16 | 14
Constipation (Gastrointestinal disorders) | 14 | 17
Diarrhoea (Gastrointestinal disorders) | 48 | 54
Dyspepsia (Gastrointestinal disorders) | 19 | 21
Nausea (Gastrointestinal disorders) | 91 | 119
Vomiting (Gastrointestinal disorders) | 41 | 49
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 16
Fatigue (General disorders) | 16 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.